CLINICAL TRIAL: NCT03606772
Title: Gynecological Presentations and Pelvic Symptoms Following Supracervical Hysterectomy for Benign Pathologies: A Survey Study
Brief Title: Gynecological Presentations Following Supracervical Hysterectomy
Acronym: GPH
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Lecturer, Tanta University
Other Study IDs: GPHysterectomy
Record Dates: First submitted 2018-07-22; First posted 2018-07-31 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Gynecological Survey

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- supracervical hysterectomy: Patients operated abdominal by removal of uterus, with removal of tubes and ovaries and retaining of cervix
  Interventions: Other: Questionanniare

INTERVENTIONS:
Other: Questionanniare — Filling printed questionnaire + Pelvic examination
  Other Names: Pelvic examination

SUMMARY:
Supracervical hysterectomy is widely common and had many complications either immediate or delayed. In these patients bleeding, infection, chronic pelvic pain are common. In these patients cervical biopsy will be done and histopathological examinations will be done to evaluate the pathology in these patients.

DETAILED DESCRIPTION:
* Study design and settings: Cross sectional descriptive studies
* Patients: 130 patients with hysterectomy recruited at Tanta University Hospital, gynecology clinics in central hospitals in Gharbia governorate will be recruited according inclusion and exclusion criteria. Inclusion criteria include all symptomatizing patients following supracervical hysterectomy, of any age, of any complaints. The
* Methods: All patients' demographic data, history, indication of hysterectomy, duration since operation, postoperative complications and their main complaint.

ELIGIBILITY:
Inclusion Criteria:

* Hysterectomy for benign pathologies

Exclusion Criteria:

* Hysterectomy for malignancy

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — ID cards
Study Population: • Patients: 1280 patients with hysterectomy recruited at Tanta University Hospital, gynecology clinics in central hospitals in Gharbia governorate
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
number of participant with gynecological symptoms following hysterectomy | 6 months
  Symptoms occurring after hysterectomy

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Dawood, Principal Investigator — Lecturer at Tanta University
Locations (1):
- Ayman Shehata Dawood, Tanta, Algharbia, Egypt

IPD SHARING:
Plan to Share IPD: No
Patients data are not allowed to be public